CLINICAL TRIAL: NCT07092202
Title: Exploratory Clinical Study on Dynamic Monitoring of cfDNA in Cerebrospinal Fluid and Peripheral Blood Using High-dose Firmonertinib Combined With Intrathecal Injection of Pemetrexed for the Treatment of EGFR Mutant NSCLC With Leptomeningeal Metastases
Brief Title: Firmonertinib Combined With Intrathecal Injection for the Treatment of EGFR Mutant NSCLC With Leptomeningeal Metastases
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTO-20240928
Record Dates: First submitted 2025-07-14; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Leptomeningeal Metastasis; NSCLC; Intrathecal Chemotherapy; Tyrosine Kinase Inhibitor
Keywords: Leptomeningeal metastasis; NSCLC; Intrathecal Chemotherapy; Firmonertinib; Tyrosine Kinase Inhibitor; cfDNA
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Firm-ITp (Experimental): 1. Firmonertinib 160mg po qd;
  2. Intrathecal injection of pemetrexed. Weight above 50kg: Induction period: 40mg/time, d1, d5 (q3w, x 4 cycles); Consolidation period: 40mg/time, q4w (pause when cerebrospinal fluid ctDNA is negative); Weight below 50kg: Induction period: 30mg/time, d1, d5 (q3w, x 4 cycles); Consolidation period: 30mg/time, q4w (pause when cerebrospinal fluid ctDNA is negative).
  Interventions: Drug: Firmonertinib; Drug: Intrathecal injection of pemetrexed

INTERVENTIONS:
Drug: Firmonertinib — Firmonertinib 160mg po qd
Drug: Intrathecal injection of pemetrexed — Intrathecal injection of pemetrexed. Weight above 50kg: Induction period: 40mg/time, d1, d5 (q3w, x 4 cycles); Consolidation period: 40mg/time, q4w (pause when cerebrospinal fluid ctDNA is negative); Weight below 50kg: Induction period: 30mg/time, d1, d5 (q3w, x 4 cycles); Consolidation period: 30mg/time, q4w (pause when cerebrospinal fluid ctDNA is negative)

SUMMARY:
Leptomeningeal metastases (LM) are a relatively rare site of metastasis in advanced non-small cell lung cancer (NSCLC), and LM patients have a poor prognosis. Numerous retrospective studies have reported that high-dose Firmonertinib can also effectively increase patient prognosis and have tolerable side effects, but there is a lack of prospective studies to confirm this. In addition, there are currently no good biomarkers for monitoring the efficacy of LM treatment. cfDNA testing can be used for early cancer screening, monitoring tumor progression, evaluating treatment response, and discovering drug resistance mechanisms. Due to the influence of the blood-brain barrier, the level of cfDNA in the plasma of LM patients is often very low, and the detection of cfDNA in cerebrospinal fluid (CSF) is more advantageous. Therefore, exploring the dynamic monitoring of LM treatment efficacy using CSF cfDNA is of great significance for improving patient prognosis. Based on this, the applicant intends to conduct a prospective, multicenter, single-arm, post-market exploratory clinical trial on the treatment methods and efficacy monitoring of NSCLC-LM patients. The aim was to explore whether cfDNA has the potential to become a biomarker for LM efficacy monitoring and to validate the efficacy and safety of high-dose fumatinib combined with intrathecal injection in the treatment of NSCLC-LM patients.

DETAILED DESCRIPTION:
Leptomeningeal metastases (LM) are a relatively rare site of metastasis in advanced non-small cell lung cancer (NSCLC), and LM patients have a poor prognosis. Once diagnosed, if left untreated, the overall survival (OS) is only 4-6 weeks, and the appearance of LM is often significantly associated with EGFR mutations. At present, the commonly used treatment for LM metastasis in clinical practice is systemic targeted therapy combined with local intrathecal injection of chemotherapy drugs, such as intrathecal injection of pemetrexed. The BLOOM study showed that increasing the dose of osimertinib (160mg) showed promising efficacy in advanced NSCLC patients with previous EGFR-TKI treatment failure and concomitant leptomeningeal metastasis, while double-dose targeted drugs had good safety and controllable adverse reactions. Numerous retrospective studies have reported that high-dose Firmonertinib can also effectively increase patient prognosis and have tolerable side effects, but there is a lack of prospective studies to confirm this. In addition, there are currently no good biomarkers for monitoring the efficacy of LM treatment. cfDNA testing can be used for early cancer screening, monitoring tumor progression, evaluating treatment response, and discovering drug resistance mechanisms. Due to the influence of the blood-brain barrier, the level of cfDNA in the plasma of LM patients is often very low, and the detection of cfDNA in cerebrospinal fluid (CSF) is more advantageous. Moreover, there are relatively few studies on this topic; therefore, exploring the dynamic monitoring of LM treatment efficacy using CSF cfDNA is of great significance for improving patient prognosis. Based on this, the applicant intends to conduct a prospective, multicenter, single-arm, post-market exploratory clinical trial on the treatment methods and efficacy monitoring of NSCLC-LM patients. The dynamic monitoring of cfDNA in cerebrospinal fluid and peripheral blood was used to evaluate the efficacy and safety of high-dose fumatinib combined with intrathecal injection of pemetrexed in the treatment of EGFR mutant NSCLC with leptomeningeal metastases. The aim was to explore whether cfDNA has the potential to become a biomarker for LM efficacy monitoring and to validate the efficacy and safety of high-dose fumatinib combined with intrathecal injection in the treatment of NSCLC-LM patients.

ELIGIBILITY:
Inclusion Criteria:

* Obtain an informed consent form signed by the patient or their legal representative;
* Age greater than or equal to 18 years old;
* According to the 9th edition TNM staging of lung cancer by the International Association for the Study of Lung Cancer and the Joint Committee on Cancer Staging in the United States, metastatic (stage IV) NSCLC with histological or cytological confirmation;
* Confirmed by histological or cytological specimens tested in the central laboratory to have EGFR exon 19 deletion mutation (19DEL) or exon 21 L858R point mutation (L858R), which can exist alone or in combination;
* ECOG physical condition score is 0-3 points, with an expected life expectancy of ≥ 12 weeks;
* According to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1), there should be at least one measurable lesion;
* According to the "EANO-ESMO" diagnostic criteria for meningeal metastasis (Type I: positive cerebrospinal fluid cytology or biopsy; Type II: limited to typical clinical symptoms and neuroimaging findings), for clinical judgment. Patients with leptomeningeal metastases who can be included in the study are type I patients and type II patients with EGFR mutations in cerebrospinal fluid ctDNA; merged brain parenchymal metastases can also be included in the study;
* Progress in first-line treatment with first and second-generation EGFR-TKI;
* Progress in first-line conventional dose treatment with third-generation EGFR-TKI;
* The subject must accept and be able to cooperate with the lumbar puncture procedure, and confirm that there are no contraindications to chemotherapy or lumbar puncture;
* At least 4 weeks before treatment, all extracranial symptoms must be stable, and there must be no CNS complications requiring emergency neurosurgical intervention.

Exclusion Criteria:

* Squamous cell carcinoma of the lung;
* Known history of hypersensitivity reactions to drugs with or without active excipients or similar structures or categories to the investigational drug for famotinib/pemetrexed;
* Confirmed EGFR exon 20 insertion mutation;
* At the beginning of drug treatment, if the toxicity associated with previous anti-tumor therapy has not recovered to ≤ CTCAE Grade 1, except for peripheral neurotoxicity caused by hair loss or chemotherapy ≤ CTCAE Grade 2;
* Excluding skin basal cell carcinoma, cervical carcinoma in situ, and ductal carcinoma of the breast that have been effectively controlled and have been diagnosed with other malignant tumors or have a history of other malignant tumors in the past 5 years;
* Patients who are deemed ineligible by researchers to participate in this study, such as those who are highly likely to be unable to comply with the study protocol, constraints, and requirements, or other situations determined by the researcher at their discretion;
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  From the date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Dong, Dr, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chemi F, Pearce SP, Clipson A, Hill SM, Conway AM, Richardson SA, Kamieniecka K, Caeser R, White DJ, Mohan S, Foy V, Simpson KL, Galvin M, Frese KK, Priest L, Egger J, Kerr A, Massion PP, Poirier JT, Brady G, Blackhall F, Rothwell DG, Rudin CM, Dive C. cfDNA methylome profiling for detection and subtyping of small cell lung cancers. Nat Cancer. 2022 Oct;3(10):1260-1270. doi: 10.1038/s43018-022-00415-9. Epub 2022 Aug 8. PMID 35941262
- [Background] Yan W, Liu Y, Li J, Han A, Kong L, Yu J, Zhu H. Whole brain radiation therapy does not improve the overall survival of EGFR-mutant NSCLC patients with leptomeningeal metastasis. Radiat Oncol. 2019 Sep 14;14(1):168. doi: 10.1186/s13014-019-1376-z. PMID 31521171
- [Background] Fan C, Jiang Z, Teng C, Song X, Li L, Shen W, Jiang Q, Huang D, Lv Y, Du L, Wang G, Hu Y, Man S, Zhang Z, Gao N, Wang F, Shi T, Xin T. Efficacy and safety of intrathecal pemetrexed for TKI-failed leptomeningeal metastases from EGFR+ NSCLC: an expanded, single-arm, phase II clinical trial. ESMO Open. 2024 Apr;9(4):102384. doi: 10.1016/j.esmoop.2024.102384. Epub 2024 Feb 19. PMID 38377785
- [Background] Fan C, Zhao Q, Li L, Shen W, Du Y, Teng C, Gao F, Song X, Jiang Q, Huang D, Jin Y, Lv Y, Wei L, Shi T, Zhao X, Gao N, Jiang Z, Xin T. Efficacy and Safety of Intrathecal Pemetrexed Combined With Dexamethasone for Treating Tyrosine Kinase Inhibitor-Failed Leptomeningeal Metastases From EGFR-Mutant NSCLC-a Prospective, Open-Label, Single-Arm Phase 1/2 Clinical Trial (Unique Identifier: ChiCTR1800016615). J Thorac Oncol. 2021 Aug;16(8):1359-1368. doi: 10.1016/j.jtho.2021.04.018. Epub 2021 May 11. PMID 33989780
- [Background] Qi R, Fu X, Yu Y, Xu H, Shen M, He S, Lv D. Efficacy and safety of re-challenging 160 mg furmonertinib for advanced NSCLC after resistance to third-generation EGFR-TKIs targeted agents: A real-world study. Lung Cancer. 2023 Oct;184:107346. doi: 10.1016/j.lungcan.2023.107346. Epub 2023 Aug 17. PMID 37604026
- [Background] Cheng D, Tang S, Li D, Zhao W, Wei W, Fang C, Ji M. Successful salvage therapy using high-dose furmonertinib (AST2818) for non-small-cell lung cancer after Osimertinib resistance: a case report. Anticancer Drugs. 2022 Sep 1;33(8):768-772. doi: 10.1097/CAD.0000000000001368. Epub 2022 Aug 10. PMID 35946524
- [Background] Xu Z, Hao X, Wang Q, Yang K, Li J, Xing P. Intracranial efficacy and safety of furmonertinib 160 mg with or without anti-angiogenic agent in advanced NSCLC patients with BM/LM as salvage therapy. BMC Cancer. 2023 Mar 4;23(1):206. doi: 10.1186/s12885-023-10676-x. PMID 36870951
- [Background] Shi Y, Hu X, Zhang S, Lv D, Wu L, Yu Q, Zhang Y, Liu L, Wang X, Cheng Y, Ma Z, Niu H, Wang D, Feng J, Huang C, Liu C, Zhao H, Li J, Zhang X, Jiang Y, Gu C. Efficacy, safety, and genetic analysis of furmonertinib (AST2818) in patients with EGFR T790M mutated non-small-cell lung cancer: a phase 2b, multicentre, single-arm, open-label study. Lancet Respir Med. 2021 Aug;9(8):829-839. doi: 10.1016/S2213-2600(20)30455-0. Epub 2021 Mar 26. PMID 33780662
- [Background] Yang JCH, Kim SW, Kim DW, Lee JS, Cho BC, Ahn JS, Lee DH, Kim TM, Goldman JW, Natale RB, Brown AP, Collins B, Chmielecki J, Vishwanathan K, Mendoza-Naranjo A, Ahn MJ. Osimertinib in Patients With Epidermal Growth Factor Receptor Mutation-Positive Non-Small-Cell Lung Cancer and Leptomeningeal Metastases: The BLOOM Study. J Clin Oncol. 2020 Feb 20;38(6):538-547. doi: 10.1200/JCO.19.00457. Epub 2019 Dec 6. PMID 31809241
- [Background] Lee J, Choi Y, Han J, Park S, Jung HA, Su JM, Lee SH, Ahn JS, Park K, Ahn MJ. Osimertinib Improves Overall Survival in Patients With EGFR-Mutated NSCLC With Leptomeningeal Metastases Regardless of T790M Mutational Status. J Thorac Oncol. 2020 Nov;15(11):1758-1766. doi: 10.1016/j.jtho.2020.06.018. Epub 2020 Jul 9. PMID 32652216
- [Background] Kawamura T, Hata A, Takeshita J, Fujita S, Hayashi M, Tomii K, Katakami N. High-dose erlotinib for refractory leptomeningeal metastases after failure of standard-dose EGFR-TKIs. Cancer Chemother Pharmacol. 2015 Jun;75(6):1261-6. doi: 10.1007/s00280-015-2759-y. Epub 2015 Apr 29. PMID 25921002
- [Background] Jackman DM, Cioffredi LA, Jacobs L, Sharmeen F, Morse LK, Lucca J, Plotkin SR, Marcoux PJ, Rabin MS, Lynch TJ, Johnson BE, Kesari S. A phase I trial of high dose gefitinib for patients with leptomeningeal metastases from non-small cell lung cancer. Oncotarget. 2015 Feb 28;6(6):4527-36. doi: 10.18632/oncotarget.2886. PMID 25784657
- [Background] Le Rhun E, Weller M, van den Bent M, Brandsma D, Furtner J, Ruda R, Schadendorf D, Seoane J, Tonn JC, Wesseling P, Wick W, Minniti G, Peters S, Curigliano G, Preusser M; EANO Guidelines Committee and ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Leptomeningeal metastasis from solid tumours: EANO-ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. ESMO Open. 2023 Oct;8(5):101624. doi: 10.1016/j.esmoop.2023.101624. Epub 2023 Sep 19. PMID 37863528
- [Background] Wilcox JA, Chukwueke UN, Ahn MJ, Aizer AA, Bale TA, Brandsma D, Brastianos PK, Chang S, Daras M, Forsyth P, Garzia L, Glantz M, Oliva ICG, Kumthekar P, Le Rhun E, Nagpal S, O'Brien B, Pentsova E, Lee EQ, Remsik J, Ruda R, Smalley I, Taylor MD, Weller M, Wefel J, Yang JT, Young RJ, Wen PY, Boire AA. Leptomeningeal metastases from solid tumors: A Society for Neuro-Oncology and American Society of Clinical Oncology consensus review on clinical management and future directions. Neuro Oncol. 2024 Oct 3;26(10):1781-1804. doi: 10.1093/neuonc/noae103. PMID 38902944